CLINICAL TRIAL: NCT01320254
Title: Panitumumab in Combination With Cisplatin/Gemcitabine Chemotherapy in Patients With Cholangiocarcinomas - a Randomized Clinical Phase II Study
Brief Title: PiCCA Study (Panitumumab in Combination With Cisplatin/Gemcitabine)
Acronym: PiCCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-Nr.: 2010-018850-11
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Cholangiocarcinomas
Keywords: Palliative treatment; Panitumumab; Cisplatin; Cisplatinum; Gemcitabine; Vectibix
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cisplatin; Gemcitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin, Gemcitabine and Panitumumab (Experimental): Experimental Arm with cisplatin 25mg/sq.m. at day 1 + 8, gemcitabine 1000mg/ sq.m.at day 1 + 8 and panitumumab 9mg/kg BW at day 1. Cycle will be repeated every 3 weeks.
  Interventions: Drug: Cisplatin, Gemcitabine, Panitumumab
- Cisplatin and Gemcitabine (Active Comparator): Cisplatin 25mg/sq.m. at day 1 + 8 and Gemcitabine 1000 mg/sq.m. at day 1 + 8. Cycle will be repeated every 3 weeks.
  Interventions: Drug: Cisplatin, Gemcitabine

INTERVENTIONS:
Drug: Cisplatin, Gemcitabine, Panitumumab — Cisplatin 25mq/sq.m. at day 1+8 and Gemcitabine 1000mg/sq.m. at day 1 + 8 Panitumumab 9mg/kg BW at day 1
  Other Names: Vectibix (Panitumumab); Gemzar (Gemcitabine); Cisplatin 0.5mg/ml solution medac (Cisplatin)
  Arms: Cisplatin, Gemcitabine and Panitumumab
Drug: Cisplatin, Gemcitabine — Cisplatin 25mq/sq.m. at day 1+8 and Gemcitabine 1000mg/sq.m. at day 1 + 8
  Other Names: Gemzar (Gemcitabine); Cisplatin 0.5mg/ml solution medac (Cisplatin)
  Arms: Cisplatin and Gemcitabine

SUMMARY:
The purpose of this study is to determine the efficacy of panitumumab plus cisplatin/gemcitabine (CisGem) combination chemotherapy in KRAS wild-type biliary tract cancer patients without systemic pre-treatment, compared to the historical data and to the randomised control group without the antibody, which verifies the historically based assumption.

DETAILED DESCRIPTION:
The rationale of the study is the assessment of the clinical activity of Panitumumab in conjunction with standard Cisplatin/Gemcitabine chemotherapy in patients with cholangiocarcinomas and gall bladder carcinomas in 1st-line therapy.

Cholangiocarcinoma (CCA) is an epithelial cancer originating from the bile ducts with features of cholangiocyte differentiation. CCA is the second most common primary hepatic malignancy, and epidemiologic studies suggest its incidence is increasing in Western countries. Hepatobiliary malignancies account for 13% of the 7.6 million annual cancer-related deaths worldwide and CCA accounts for approximately 20% of the deaths from hepatobiliary malignancies (Kubicka and Manns 2000; Kubicka 2004; Blechacz and Gores 2008; Malek et al. 2007).

The only curative option for patients with gallbladder- or bile duct cancer is surgical resection. Advanced CCA has a devastating prognosis. There are only limited numbers of studies about the systemic treatment options for biliary cancers. Gallbladder and bile duct carcinomas are moderately chemotherapy-sensitive tumors. The objective response rates in phase II studies with 5-FU or gemcitabine monochemotherapy are between 10 - 30 % (Kubicka et al. 2001b). Higher response rates between 20 - 50 % have been observed in phase II studies with combination chemotherapy, in particular with the combination of gemcitabine/cisplatin (Kubicka 2004; Malek et al. 2007).

Recently for the first time an improvement of overall survival has been demonstrated in a large randomized phase III trial with chemotherapy combination of cisplatin and gemcitabine (n=206) compared to gemcitabine mono-chemotherapy (n=204) (Valle et al. 2009). Median overall survival was 8,2 month in the monotherapy arm versus 11,7 month in the combination arm (p=0.002). As a consequence of this study the combination of Cisplatin (25mg/m² d1,8) and Gemcitabine (1000mg/m² d1,8) should be considered as the standard first line chemotherapy for patients with irresectable cholangio- or gallbladder carcinomas.

The growing understanding of the molecular pathogenesis of CCA opens new therapeutic options for molecular targeting (Blechacz and Gores 2008). In particular EGFR signaling appears to be important for tumor growth of CCA. Inhibition of EGFR signaling has been shown to significantly suppress CCA cell growth (Blechacz and Gores 2008). In addition EGFR can directly be activated by bile acids and promote CCA cell proliferation, a potential explanation for the tropism exerted by CCA for the biliary tree. It has been shown that EGFR activation is sustained in CCA by failure to internalize the ligand-receptor complex, a homeostatic mechanism essential for receptor inactivation. EGFR phosphorylation results in activation of the downstream kinases p42/44 MAPK and p38 MAPK, which in turn increase cyclooxygenase 2 expression in CCA cells.

Further evidence for the essential contribution of EGFR-signalling comes from studies with IL-6 (Blechacz and Gores 2008). IL-6 is a key cytokine in the pathogenesis of CCA. IL-6 is produced at high levels by CCA cells, and elevated IL-6 serum concentrations have been reported in CCA patients. It has been shown that there is a cross-communication between IL-6 and EGFR resulting in IL-6 mediated overexpression of EGFR.

Recently the first results of a randomized phase II study of gemcitabine and oxaliplatin (GEMOX) alone or in combination with cetuximab in patients with advanced biliary cancer have been reported (Malka et al. 2009). The primary objective of the study was a 4-month PFS rate of more than 60% in the experimental arm with cetuximab. The included patients were not monitored for RAS or B-RAF mutations. However compared to GEMOX chemotherapy (n=51), GEMOX+cetuximab (n=50) showed an increased 4-month PFS-rate (50% versus 61%) and an improved median PFS (5 versus 7 months). This is the first evidence from a randomized trial that anti-EGFR therapy may be effective for patients with cholangiocarcinomas and gallbladder carcinomas.

KRAS is a downstream molecule in the EGFR-pathway. Recently it has been shown that oncogenic RAS mutations are predictive for poor efficacy of an anti-EGFR-therapy in colorectal cancer. Conversely patients with colorectal cancers harbouring KRAS wild-type showed frequently dramatic tumor responses upon anti-EGFR-treatment, indicating that colorectal cancers with KRAS wild type are highly susceptible for an anti-EGFR-therapy. Although dysregulation of KRAS is commonly observed in malignancies, mutations of KRAS have only been described in 12% to 54% of intrahepatic CCA (Kubicka et al. 2001a; Blechacz and Gores 2008, Gruenberger et al 2009). This is in sharp contrast to pancreatic ductal carcinoma where KRAS mutations are present in approximately 90% of cancers. Thus, despite shared developmental ontology between the pancreatic ducts and the biliary tree, their adult cancers are different and may explain the negative result of a phase III studies in pancreatic cancer with Cetuximab (anti-EGFR-antibody).

Very preliminary and sparse data from a recent small phase II study with cetuximab do not allow to speculate whether the RAS status does predict the response in cholangiocarcinomas similarly to colorectal cancers (Gruenberger et al. 2009). However, due to the clear evidence of absence of efficacy in mutant KRAS colorectal cancer, the presumptive population "enrichment" should be applied in this first trial on biliary duct cancer, which is to focus on KRAS wild type patients.

Since most of the patients with CCA are treated in large centers a chemotherapy protocol with limited numbers of intravenous infusions appears to be very comfortable for patients with CCA. A further argument for the investigation of Cisplatin/Gemcitabine/Panitumumab in a randomized phase II study is the fact that the 3-week interval of the Cis/Gem protocol fits very well into the 3-week interval of the Panitumumab schedule.

ELIGIBILITY:
Inclusion Criteria:

* Signed,dated informed consent before start of specific protocol procedures
* Histologically/cytologically documented diagnosis of cholangiocarcinoma or gall bladder carcinoma
* At least one measurable site of disease following RECIST V. 1.1 criteria
* Wild-type KRAS status as assessed by standardized PCR
* Unresectable, locally advanced or metastatic disease
* Age > 18 years old
* ECOG Performance Status 0 or 1
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver (with stenting for any obstruction, if required) and renal function (lab. assessment within 7 days prior to screening):
* Hemoglobin > 10.0 g/dl
* Leukocyte count > 3.000/mm3 ; absolute neutrophil count (ANC) > 1.500/mm3
* Platelet count 100.000/mm³
* Total bilirubin < 5,0 times the upper limit of normal
* ALT and AST < 3 x upper limit of normal
* Alkaline phosphatase < 5 x ULN
* PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
* Serum creatinine < 1.5 x upper limit of normal and creatinine clearance > 60 ml/min
* Magnesium ≥ lower limit of normal; calcium ≥ lower limit of normal
* The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations
* Negative pregnancy test performed within 7 days prior to the start of treatment, and willingness to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly)

Exclusion Criteria:

* KRAS mutation
* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment
* History of interstitial lung disease, e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* History of HIV infection or chronic hepatitis B
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Pre-existing neuropathy > grade 1 (NCI CTCAE), except for loss of tendon reflex (patellar tendon reflex)
* Symptomatic or known brain metastases.A scan to confirm the absence of brain metastases is not required -Patients with seizure disorder requiring medication (such as steroids or anti- epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Patients with second primary cancer,except adequately treated basal skin cancer or carcinoma in-situ of the cervix
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
* No prior anti-cancer chemotherapy,radiotherapy(excluding palliative radiotherapy administered more than 4 weeks prior to study entry),endocrine or immunotherapy
* Investigational drug therapy outside of this trial during or within 4weeks of study entry
* Major surgery within 4 weeks of starting the study and patients must have recovered from effects of major surgery
* Prior anti-EGFR therapy
* Autologous bone marrow transplant or stem cell rescue within 4 months of study
* Breast-feeding patients
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's understanding of the informed consent procedure, participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-06; Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
progression-free survival rate | 6 months
  The progression-free survival rate at six months (primary endpoint) is defined as the number of patients recorded to be free of progression (according to RECIST) at this time point, divided by the number of patients randomized to the respective arm.

SECONDARY OUTCOMES:
Tumor response | 48 weeks
  Tumor response according to RECIST criteria within the first 48 weeks of treatment
Progression-free survival | 3 years
  Progression-free survival (PFS) will be defined as the time from randomisation to the time of disease progression or relapse (according to RECIST) or death, or to the date of last assessment without any such event (censored observation).
Overall survival | 3 years
  The duration of overall survival (OS) will be determined by measuring the time interval from randomisastion to the date of death or last observation (censored).
Number of Participants with Adverse Events as a Measure of Toxicity/Safety | 3 years
Translational research | 3 years
  assessment/ correlation of tumor response with KRAS (mandatory)
  alterations in cholangiocarcinomas and gallbladder cancer (EGFR, PTEN, BRAF)through optional translational research

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Vogel, PD Dr. MD, Study Chair — Hannover Medical School
Locations (16):
- Germany (16):
  - Esslingen Hospital, Esslingen am Neckar, Baden-Wurttemberg
  - University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - National Centre for Tumor Diseases (NCT), Heidelberg, Baden-Wurttemberg
  - University Hospital Mannheim, Mannheim, Baden-Wurttemberg
  - Kreiskliniken Reutlingen GmbH, Reutlingen, Baden-Wurttemberg
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - Klinikum rechts der Isar der TU München, München, Bavaria
  - University Hospital Regensburg, Regensburg, Bavaria
  - Charité Berlin, Berlin, Berlin-City
  - University Hospital Hamburg-Eppendorf, Hamburg, Free City of Hamburg
  - University Hospital Marburg, Marburg, Hesse
  - Medical School Hannover, Hanover, Lower Saxony
  - University Hospital Köln, Cologne, Northrhine-Westfalia
  - University Hospital Essen, Essen, Northrhine-Westfalia
  - University Hospital Mainz, Mainz, Rhineland-Palatinate
  - Magdeburg Hospital, Magdeburg, Saxony-Anhalt

REFERENCES:
- [Derived] Vogel A, Kasper S, Bitzer M, Block A, Sinn M, Schulze-Bergkamen H, Moehler M, Pfarr N, Endris V, Goeppert B, Merx K, Schnoy E, Siveke JT, Michl P, Waldschmidt D, Kuhlmann J, Geissler M, Kahl C, Evenkamp R, Schmidt T, Kuhlmann A, Weichert W, Kubicka S. PICCA study: panitumumab in combination with cisplatin/gemcitabine chemotherapy in KRAS wild-type patients with biliary cancer-a randomised biomarker-driven clinical phase II AIO study. Eur J Cancer. 2018 Mar;92:11-19. doi: 10.1016/j.ejca.2017.12.028. Epub 2018 Feb 3. PMID 29413685